CLINICAL TRIAL: NCT01742663
Title: A Randomized, Double-Blind, Multiple-Site, Placebo-Controlled, Parallel Design Study Comparing Diclofenac Sodium Gel 3% (Taro Pharmaceuticals Inc.) to Solaraze® (Diclofenac Sodium) Gel 3% (Fougera Pharms) in the Treatment of Actinic Keratosis.
Brief Title: A Study Comparing Diclofenac Sodium Gel 3% to Solaraze® Gel 3% in the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCSG 1213
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Actinic Keratosis
Keywords: Diclofenac Sodium Gel 3%; Solaraze® (diclofenac sodium) Gel 3%; Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diclofenac Sodium Gel 3% (Experimental): Diclofenac Sodium Gel 3% (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Diclofenac Sodium Gel 3%
- Solaraze® (diclofenac sodium) Gel 3% (Active Comparator): Solaraze® (diclofenac sodium) Gel 3% (Fougera Pharms)
  Interventions: Drug: Solaraze® (diclofenac sodium) Gel 3%
- Vehicle Topical Gel (Placebo Comparator): Vehicle Topical Gel (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Vehicle Topical Gel

INTERVENTIONS:
Drug: Diclofenac Sodium Gel 3% — Diclofenac Sodium Gel 3% (Taro Pharmaceuticals Inc.) applied twice daily for 60 days.
  Arms: Diclofenac Sodium Gel 3%
Drug: Solaraze® (diclofenac sodium) Gel 3% — Solaraze® (diclofenac sodium) Gel 3% (Fougera Pharms)applied twice daily for 60 days.
  Arms: Solaraze® (diclofenac sodium) Gel 3%
Drug: Vehicle Topical Gel — Vehicle Topical Gel (Taro Pharmaceuticals Inc.) applied twice daily for 60 days.
  Arms: Vehicle Topical Gel

SUMMARY:
The objective of this study is to compare the relative efficacy and safety of the test formulation diclofenac sodium gel 3% (Taro Pharmaceuticals Inc.) to the marketed formulation Solaraze® (diclofenac sodium) Gel 3% (Fougera Pharms) in the treatment of actinic keratosis.

Both the test and reference formulations will also be compared to a placebo formulation to test for superiority.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Immunocompetent male or non-pregnant, non-lactating female at least 18 years of age.
* Diagnosis of AK with at least 5 and no more than 10 clinically typical, visable, discrete, nonhyperkeratotic, nonhypertrophic AK lesions each at least 4 mm in diameter on the face and/or bald scalp contained within a 25 cm2 treatment area.
* Women either must be 1 year post-menopausal, surgically sterile, or if they are of child-bearing potential they must have been using systemic birth control, IUD or Norplant for at least 28 days prior to treatment start, or used barrier methods consistently at least 14 days before study gel administration, had a normal menstrual cycle for the month prior to the start of treatment, have a negative urine pregnancy test result upon entry into the study and agree to use a medically accepted form of birth control throughout the study period.
* Free from any systemic or dermatologic disorder that, in the opinion of the investigator, will interfere with the study results or increase the risks of AEs.
* Any skin type or race, providing the skin pigmentation will allow discernment of erythema.
* Willingness and capability to cooperate to the extent and degree required by the protocol.

Exclusion Criteria:

* Active gastrointestinal ulceration or bleeding.
* Current or history of severe renal or hepatic impairment.
* Presence of atopic dermatitis, basal cell carcinoma, squamous cell carcinoma, eczema, psoriasis, rosacea, sunburn or other possible confounding skin conditions on the face or bald scalp.
* Use within six months prior to randomization of oral isotretinoin.
* Use within six months prior to baseline on the face or bald scalp of chemical peel, dermabrasion, laser abrasion, PUVA therapy or UVB therapy.
* Use within one month prior to baseline on the face or bald scalp of cryodestruction or chemodestruction, curettage, photodynamic therapy, surgical excision, topical 5-fluorouracil, topical corticosteroids, topical diclofenac, topical Imiquimod, topical retinoids or other treatments for actinic keratosis including glycolic acids or over-the-counter products containing retinol, alpha or beta hydroxy acids.
* Use within one month prior to baseline of immunomodulators or immunosuppressive therapies, interferon, systemic corticosteroids or cytotoxic drugs.
* Known allergies to diclofenac sodium, benzyl alcohol, polyethylene glycol monomethyl ether 359, hyaluronate sodium or any excipients in the test or reference gels.
* Receiving 5-Fluorouracil or other systemic cancer chemotherapy within 6 months prior to study entry.
* Any condition, medical, psychological or social, that, in the investigator's opinion, would interfere with participation in the study.
* Women who are pregnant or planning pregnancy or lactating during the study.
* Participation in any investigational drug study within 30 days of enrollment or previous participation in this study.
* Employees or family members of employees of the research center or investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Study day 90 (30 days after completion of 60 days of treatment)
  Bioequivalence will be determined by evaluating the proportion of patients in the test and reference groups with 100% clearance of all AK lesions in the treatment area.

SECONDARY OUTCOMES:
Superiority to placebo | Study day 90 (30 days after completion of 60 days of treatment)
  The superiority of the test and reference gels against the placebo will be tested by the proportion of patients showing 100% clearance of actinic keratosis lesions at Day 90 (30 days after completion of 60 days of treatment)using the modified intent to treat population and last observation carried forward.